CLINICAL TRIAL: NCT01953939
Title: PhD Research Project: Clinimetric Properties of Outcome Measures of Physical Function Used With Lower Limb Amputees, Study 2
Brief Title: Outcome Measures for Lower Limb Amputees - A Repeatability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Judy Scopes, PhD Student, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: QMU/JS0122
Record Dates: First submitted 2013-09-16; First posted 2013-10-01 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Lower Limb Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prosthetic Limb Users (Experimental): Single lower limb amputees who are wearing their artificial limb all day and are using them outdoors for the majority of the time will be enrolled into this reliability study.
  Interventions: Other: Prosthetic Limb Users

INTERVENTIONS:
Other: Prosthetic Limb Users — There will be a time period of 7-10 days between data collection visits in this test-retest study which is measuring reliability in the functional outcome measures regularly used in clinical practice.

SUMMARY:
During any period of rehabilitation it is important to select meaningful tests that; measure what you want, are responsive to changes in the patient's condition and, easy to use in the clinical settings. With an amputee such tests may help make sure that rehabilitation programmes and the prosthesis (artificial leg) provided are tailored for the individual. New prosthetic technology is continually being developed and the active amputee now demands more from their artificial limbs. Making sure that they get the right rehabilitation programmes and the most appropriate prosthesis will help them perform to their best.

Twenty lower limb amputees who have had their artificial limb for at least one year will be recruited into this study. They will be asked to complete 2 walking tests and 4 questionnaires that measure different aspects of their condition from the comfort of the socket to their perceived ability to undertake everyday tasks. Each of the tests give a score or grade which represents the level of their ability, as judged by the test, at that given time point. The tests will be repeated on a second occasion between seven to ten days after the first.

By measuring the changes in the scores on these two occasions it is hoped that indices of reliability can be established for these particular tests that have been shown to be most widely used by Health Professional involved in the rehabilitation of amputees across the UK. It is also hoped that the minimal detectable change (MDC) can also be calculated for these tests. By understanding the MDC for a test then anyone using it will be able to know whether any changes in scores detected are real changes due to changes in the patient's abilities or just down to chance.

DETAILED DESCRIPTION:
The Outcome Measures (tests) to be used in this study were identified from a survey of Health Professionals across the UK. The top 5 in use were:

SIGAM Mobility Grades The Special Interest Group in Amputee Medicine (SIGAM) Mobility Grades describe a single-item scale of amputee mobility. A self-reported questionnaire has 21 yes/no items and when the answers are applied to an algorithm a final grade is assigned. There are 8 grades that can be assigned.

Timed up and go (TUAG) The TUAG test is a standardised quantitative measure of most of the manoeuvres required for 'basic mobility'. The subject is timed as they stand up from a chair, walk 3m, turn and return to the chair. The score is the time, in seconds, taken to complete the circuit.

2 Minute Walk Test A timed walk test is often used to measure functional exercise capacity. Participants are instructed to walk from end to end of an enclosed quiet corridor, covering as much ground as possible in two minutes. The score will be the distance walked in metres.

Locomotor Capability Index LCI-5) The Locomotor Capability Index (LCI-5) is a self-administered scale specifically designed for use with lower limb amputees. It has 14 questions about locomotor activities. The answers required are either yes or no to questions phrased such as: "Would you say you are able to do the following activities with your prosthesis on?" The total scores from each activity are totalled for a possible maximum score of 56.

Socket Comfort Score This score is a subjective measure of how comfortable the amputee feels the socket is at the time the score is taken. Amputees are asked a standard question: 'On a 0 - 10 scale, if 0 represents the most uncomfortable socket fit you can imagine, and 10 represents the most comfortable socket fit, how would you score the comfort of the socket fit of your artificial limb at the moment?" Their response on the 11 point scale is then recorded.

Finally the EQ-5D™ will be administered. The EQ-5D™ is a self-administered, standardised instrument that measures health outcomes. It provides a simple descriptive profile and a single index for the participants health status at the time of the test.

At the first Test Visit (TV1) written consent will be obtained from the amputee by the Researcher and the amputee will be enrolled as a study participant. Baseline measurements for all the tests will also be taken at this visit as well as basic demographic data recording age, cause of amputation, level of amputation and any relevant concomitant medical history.

This study utilises a test-retest methodology and Test Visit 2 (TV2) will occur within 7 and 10 days of TV1 when the tests will be repeated.

Every effort will be made to complete the tests at the same time of day for each of the participant's study visits and the order of the measurements will be randomly assigned at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Single lower limb amputee, at either trans-tibial or trans-femoral level
* Aged 18 years or older
* Using a prosthesis (artificial limb) for at least 1 year
* Wearing their artificial limb at least 8 hours per day
* Has the ability to walk over different surfaces outdoors, i.e. is an active-user outdoors

Exclusion criteria:

* Any recent (within 3 months) changes of prosthetic components or physiotherapy treatment.
* Any co-morbidities that prevent the participant undertaking any of the physical activities involved in the OMs
* Poor cognition as identified by the patient's clinical team, which may prevent the patient from fully understanding the written questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reliability of functional outcome measures | 1 week
  The scores of all the Outcome Measures under investigation will be noted at Test Visit 1(TV1) and then on a second occasion, 7 to 10 days later, at Test Visit 2 (TV2). Test-retest reliability using the Intraclass Correlation Coefficient and Bland Altman limit of agreements will be calculated for each of the Outcome Measures.

SECONDARY OUTCOMES:
Minimal detectable change (MDC) of functional OMs | 1 week
  The individual differences in the scores of each of the Outcome Measures between Test Visit 1(TV1) and a second occasion 7 to 10 days later , at Test Visit 2 (TV2) will be calculated. The standard error of measurement (SEM) will then be used to calculate the minimal detectable change (MDC), with a 90% confidence interval, for each of the Outcome Measures.

CONTACTS AND LOCATIONS:
Overall Officials: Marietta van der Linden, MSc, PhD, Study Director — Queen Margaret University, Edinburgh, UK; Judy Scopes, MPhil, Principal Investigator — Queen Margaret University, Edinburgh, UK
Locations (1):
- Astley Ainslie Hospital, Edinburgh, United Kingdom